CLINICAL TRIAL: NCT02568280
Title: A Randomised Trial Investigating the Postprandial Glucose Metabolism After Treatment With Faster-acting Insulin Aspart in Subjects With Type 1 Diabetes
Brief Title: Investigating the Postprandial Glucose Metabolism After Treatment With Faster-acting Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3922; 2014-004144-35 (EudraCT Number); U1111-1162-2053 (Other: WHO)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Faster aspart (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Insulin aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Administered subcutaneously (S.C., under the skin).Subjects will be individually dosed.
  Arms: Faster aspart
Drug: insulin aspart — Administered subcutaneously (S.C., under the skin).Subjects will be individually dosed.
  Arms: Insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the postprandial glucose metabolism after treatment with faster-acting insulin aspart in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-64 years (both inclusive) at the time of signing informed consent
* Subjects diagnosed (clinically) with type 1 diabetes mellitus at least 365 days prior to the day of screening
* Body mass index 18.5-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Smoker (defined as a subject who is smoking at least five cigarettes or the equivalent per day) who is not able or willing to refrain from smoking or use of nicotine gum or transdermal nicotine patches during the inpatient period
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

PRIMARY OUTCOMES:
Mean change in plasma glucose concentration | From 0-1 hour after trial product administration

SECONDARY OUTCOMES:
Rate of endogenous glucose production | From 0-6 hours after trial product administration
Area under the serum insulin aspart concentration-time curve | From 0-6 hours after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Basu A, Pieber TR, Hansen AK, Sach-Friedl S, Erichsen L, Basu R, Haahr H. Greater early postprandial suppression of endogenous glucose production and higher initial glucose disappearance is achieved with fast-acting insulin aspart compared with insulin aspart. Diabetes Obes Metab. 2018 Jul;20(7):1615-1622. doi: 10.1111/dom.13270. Epub 2018 Mar 30. PMID 29493118
- [Result] Haahr H, Pieber TR, Mathieu C, Gondolf T, Shiramoto M, Erichsen L, Heise T. Clinical Pharmacology of Fast-Acting Insulin Aspart Versus Insulin Aspart Measured as Free or Total Insulin Aspart and the Relation to Anti-Insulin Aspart Antibody Levels in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2019 May;58(5):639-649. doi: 10.1007/s40262-018-0718-6. PMID 30402720
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com